CLINICAL TRIAL: NCT07118761
Title: Frailty Status in Hospitalized Persons: Artificial Intelligence-based Detection and Technology-assisted Home-based Empowerment (ART.I.DE.)
Brief Title: Home-based Empowerment Through Physical Exercise Assisted by Technology for Frail Patients
Acronym: ARTIDE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Collaborators: Università degli Studi di Ferrara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 189/2024/Sper/AOUFe
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-05

CONDITIONS: Frailty
Keywords: Exercise; Technology; Home-based training; Elderly; Frailty
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based technology-assisted Exercise (Experimental): Patients enrolled in this group will undergo an exercise-based intervention at home guided by the ARTIDE app. Each exercise session will encompass 8 walking minutes at home at a fixed slow speed to be repeated twice per day. Every week the speed will be slightly increased to maintain an adequate training stimulus.
  Interventions: Behavioral: Home-based walking training
- Control (No Intervention): Patients enrolled in this group will receive usual care, including traditional home rehabilitation, if needed.

INTERVENTIONS:
Behavioral: Home-based walking training — Patients enrolled in the experimental group will undergo an exercise-based intervention at home guided by a smartphone application. Each exercise session will encompass 8 walking minutes at home at a fixed slow speed to be repeated twice per day. Every week the speed will be slightly increased to maintain an adequate training stimulus.
  Arms: Home-based technology-assisted Exercise

SUMMARY:
This project, that lays in Health Ageing mission promoted by European Commission, aims to address the issue of frailty, a condition that poses the elderlies to increased vulnerability, deconditioning, and, ultimately, loss of independence. Frail people are exposed to a significant increase in mortality, hospitalizations and falls, with high burden for families and for the National Health Service (NHS). Nowadays, the detection of frailty is performed with more than 75 validated measures including questionnaires, scales and technologies. Moreover, frailty is usually not properly addressed, due to the limited resources in terms of personnel and programs in the NHS, and the frail patient is at high risk to be institutionalized and to definitely lose his functional independence. The project here proposed aims to address these topics, by combining clinical, rehabilitation, and engineering expertise in a unique team.

Indeed, the projects aims to empower the frail people with an home-based app-guided rehabilitation program. In order to easily develop a largely tested home-based walking program, we aim to design and develop an application, compatible with any device, that will enable each person to easily exercise at home just few minutes per day. Through a randomized-controlled clinical trial, we will verify the effectiveness of the rehabilitation program on frailty status, in promoting patients' independence, quality of life and ARTIDE score.

ELIGIBILITY:
Inclusion Criteria:

* Frail condition as determined by a Fried Frailty Score equal or more than 2,
* Barthel Index > 60
* Ability to ambulate also with assistance
* Ability to communicate with the research team
* Ability to use a smartphone or a tablet.

Exclusion Criteria:

* terminal illness;
* life-threatening conditions;
* absolute contraindications to exercise training (e.g. fracture);
* severe cognitive decline identified by a Mini-mental status examination < 18;
* incapability or unwillingness to provide informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2027-06-14 (Estimated); Study Completion 2028-07-14 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery | From enrollment to the end of treatment at 3 months
  This battery includes three different tests focusing on balance (side-by-side, semi-tandem and tandem position), gait speed (4-meter test) and lower-limb strength (5-time sit-to-stand test). The scale score ranges from 0 (lowest) to 12 (higher) by summing the points obtained in the three tests.

SECONDARY OUTCOMES:
Barthel Index | From enrollment to the end of treatment at 3 months
  Assess the functional independence in activities of daily living. This ordinal scale includes 10 items and provides a score ranging from 0 (total dependence) to 100 (total independence).
2-minute walking test | From enrollment to the end of treatment at 3 months
  Patients will be instructed to walk on a 20-meter corridor aiming at covering as much distance as possible in two minutes. Patients will be allowed to slow down the pace and/or stop in case of fatigue and symptoms. The total distance covered will be collected, as well the 0-10 rate of perceived exertion
Quality of life through EQ-5D-5L questionnaire | From enrollment to the end of treatment at 3 months
  The questionnaire includes five Likert-scale multiple choice questions and a visual analog scale to measure the current perception of quality of life.
Number of falls | From enrollment to 12 months
  Rate of falls will be collected by giving to the patients' caregiver (when possible) or directly to the patient a small diary to report the total number of falls experienced
All-cause hospitalizations | From enrollment to 12 months
  Number and rate of all-cause hospitalizations at 12 months. For each patient enrolled we will periodically analyzed the regional dataset to check for any recurrent hospitalization. In case of positive findings, the days elapsed from enrollment to the event will be recorded for additional analyses, as well as the reasons and the diagnoses
Survival rate | From enrollment to 12 months
  Number and rate of mortality at 12 months. For each patient enrolled we will periodically analyzed the regional dataset to check for any recurrent hospitalization. In case of positive findings, the days elapsed from enrollment to the event will be recorded for additional analyses, as well as the reasons and the diagnoses

CONTACTS AND LOCATIONS:
Locations (2):
- University Hospital of Ferrara, Ferrara, Italy
- Hospital Universitario Reina Sofia, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
The dataset generated from the study will be publicly available in a web repository
Supporting Information: Study Protocol
Time Frame: Start date: January 2026 End date: December 2028